CLINICAL TRIAL: NCT03848468
Title: Comparison Study: Ligasure Versus Conventional Hemorrhoidectomy in III and IV Degree Hemorrhoids.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Safia Zahir Ahmed, principal investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ServicesH
Record Dates: First submitted 2019-02-11; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Hemorrhoidectomy; Hemorrhoids Third Degree; Hemorrhoids Fourth Degree; Operative Time; Pain, Postoperative; Wound Healing; Return to Work
Keywords: Visual Analogue pain score; conventional Hemorrhoidectomy; Ligasure Hemorrhoidectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Hemorrhoidectomy

STUDY DESIGN:
Intervention Model Description: Covidien 5mm ligasure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CH(conventional Hemorrhoidectomy) (Active Comparator): conventional hemorrhoidectomy
  Interventions: Procedure: Hemorrhoidectomy
- LH (Ligasure Hemorrhoidectomy) (Experimental): Ligasure hemorrhoidectomy
  Interventions: Procedure: Hemorrhoidectomy

INTERVENTIONS:
Procedure: Hemorrhoidectomy — excision of 3rd and 4th degree hemorrhoids

SUMMARY:
A comparison study was performed between Ligasure and Milligan morgan hemorrhoidectomy to find out the outcome between these two techniques in 3rd and 4th degree hemorrhoids.This advance vessel sealing device is used to seal the pedicle of the vessel and does not burn the surrounding tissues , so the outcome was monitored in terms of operative time, post operative pain pain, duration of wound healing in 3 weeks and return to normal activities

DETAILED DESCRIPTION:
INTRODUCTION:

Milligan Morgan hemorrhoidectomy is conventional procedure in 3rd and 4th degree hemorrhoids but recent advances in ligasure hemorrhoidectomy have shown to produce favorable results. Comparison of these two is studied in terms of pain outcome as patient perceives, operative time, wound healing and return to normal activities.

OBJECTIVES:

To compare the outcome of ligasure hemorrhoidectomy with conventional hemorrhoidectomy in III and IV degree hemorrhoids.

STUDY DESIGN:

Randomized controlled trial

STUDY SETTING:

The study was conducted in surgical unit 1, Services hospital, Lahore.

DURATION OF STUDY:

Study was completed in six months after the approval of synopsis i.e. from 1st April 2014 to 30th September 2014.

DATA COLLECTION PROCEDURE:

After approval from hospital ethical committee, 100 patients fulfilling the inclusion criteria has been recruited from outdoor and emergency department. A detailed history had been taken including demographic data (age, address) and all patients had been clinically examined .Patients was divided in two groups randomly using random number tables. Group A: Conventional hemorrhoidectomy. Group B: Ligasure hemorrhoidectomy. Patients had been requested to sign an informed consent. They had been assured regarding confidentiality and expertise used for the procedure. All procedures have been performed by a single surgical operating team to control bias. Preoperatively operative time was noted. Post operatively pain had been assessed after 6 hours, 24 hours, and 48 hours, wound has been assessed in 2nd and 3rd postoperative week to assess epithelization and return to normal activities in days. All data had been collected and recorded on the Proforma

ELIGIBILITY:
Inclusion Criteria:

* patients with III and IV degree hemorrhoids assessed on proctoscopy had been included in this study.

Exclusion Criteria:

* Patients with permanently prolapsed hemorrhoids limited to one quadrant only and had been assessed on per rectal examination and proctoscopy
* Any other anorectal pathology on history and per rectal examination
* Previous anal surgery assessed by history and per rectal examination
* Inability to give informed consent
* ASA(American Society of Anesthesiologists) grade III/IV on detailed history, clinical examination and laboratory findings e.g. deranged hepatic and renal profile and evidence of ischemic heart disease

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
operative time | each participant was measured from the start of operation till the dressing i.e duration of 20 minutes to 60 minutes
  was measured from start of incision to the dressing in minutes
mean postoperative pain | each participant was individually assessed after operation in 6 hours,24 hours and 48 hours post-operative and changes noted in 48 hours
  on Visual analogue scale,a scale to assess the post operative pain ,8-10 as maximum pain, 5-7 as moderate pain, 2-4 minimum pain, 1-0 as no pain and change in final outcome has been assessed after 48 hours
wound healing | to assess change in the parameter in 3 weeks
  assessed in scheduled appointment every week and has been defined as complete epithelization on physical examination .Wound was graded as 1-sloughy, 2-no granulation, 3-granulation, 4-epithelizing , 5-completely epithelized
Return to work | assessed individually from the day of surgery to resume of daily activities i.e 1 to 7 days
  has been defined as day of discharge till resume of work that is patient is able to perform daily routine activities normally as before operation.

CONTACTS AND LOCATIONS:
Locations (1):
- services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided